CLINICAL TRIAL: NCT01353573
Title: A Randomized Trial of Robotic Compared to Fixed Gantry Radiosurgery for Brain Metastases
Brief Title: Robotic Compared to Fixed Gantry Radiosurgery for Brain Metastases
Acronym: TRICK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other); Juravinski Cancer Centre Foundation (Other)
Responsible Party: Dr. Jeffrey Noah Greenspoon Radiation Oncology Research Fellow, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JNG-001
Record Dates: First submitted 2011-05-10; First posted 2011-05-13 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Malignant Neoplasm to the Adult Brain
Keywords: Brain Neoplasms; Neoplasm Metastasis; Neoplasms
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Gantry Radiosurgery (Active Comparator): Single fraction radiosurgery will be prescribed using a Fixed Gantry Linear Accelerator
  Interventions: Radiation: Fixed Gantry Radiosurgery
- Robotic Radiosurgery (Experimental): Single fraction radiosurgery will be prescribed using a robotic linear accelerator
  Interventions: Radiation: Robotic Radiosurgery

INTERVENTIONS:
Radiation: Fixed Gantry Radiosurgery — Single fraction radiosurgery will be prescribed using a fixed gantry radiosurgery delivery system
  Other Names: Linear Accelerator Radiosurgery
  Arms: Fixed Gantry Radiosurgery
Radiation: Robotic Radiosurgery — Single fraction radiosurgery will be prescribed using a robotic radiosurgery system
  Other Names: CyberKnife Radiosurgery
  Arms: Robotic Radiosurgery

SUMMARY:
Radiosurgery is precisely delivered high dose radiation. It can be performed using multiple cobalt sources, a modified traditional gantry-based linear accelerator or a robotic linear accelerator. The treatment of brain metastases represents the most common indication for radiosurgery while new indications for this technology are continually being discovered. With the increasing importance of radiosurgery and the resource implications for radiotherapy programs the investigators have proposed the first direct technological comparison of robotic to linear accelerator radiosurgery for brain metastases.

DETAILED DESCRIPTION:
Radiosurgery can be performed using multiple Co-60 sources, a modified traditional gantry-based linear accelerator, or a robotic linear accelerator. Each technique has its own advantages and disadvantages. Co-60 radiosurgery has very precise target localization by using a rigid immobilization device. The requirement for rigid immobilization limits its treatments to the head and neck. Robotic radiosurgery permits precise radiation to be delivered without the requirement for rigid immobilization. Robotic radiosurgery uses real-time imagining, allowing it to track the cancer or internal structures as they move during treatment. Another advantage is that it can deliver many small beams of radiation (as many as 200) in a limited time period and can treat lesions anywhere in the body. A traditional gantry-based linear accelerator normally requires some form of immobilization and requires more time for multiple isocentre set up but can provide both radiosurgery and conventional treatments.

Brain metastases occur in up to 50% of patients with cancer. It has been reported up to 65% of patients with brain metastases will present with one to three lesions. This represents 18,000 patients in Ontario each year who would be eligible for radiosurgery as part of their management. Randomized trials have demonstrated improved palliation and overall survival when radiosurgery is added to conventional whole brain radiation therapy (WBRT). As a result the treatment of brain metastases currently represents the largest resource use for radiosurgery. During the commissioning and initial use of the first robotic radiosurgery device in Ontario (CyberKnife) the investigators became aware of its potential advantages for the treatment of brain metastases. Treatment planning time and on treatment time with robotic radiosurgery appeared to be better than with a traditional linear accelerator and patients appeared to be more comfortable with the minimal/ non-invasive immobilization required. Surprisingly, there were very little direct comparisons of robotic radiosurgery with other techniques in the literature and only one prospective randomized trial comparing two different approaches to delivering Co-60 radiosurgery was identified. Given the increasing importance of radiosurgery and the resource implications for radiation treatment programs in Ontario, this study is proposed to conduct a direct comparison of robotic to traditional linear accelerator radiosurgery for brain metastases. The primary outcome will be treatment planning and delivery time and an important secondary outcome is patient comfort. Treatment planning time will include immobilization preparation, CT simulation, image fusion, radiation planning and treatment plan quality assurance. Treatment delivery time will include patient set up, target localization and treatment delivery. The Juravinski Cancer Centre (JCC) and McMaster University are uniquely posed to perform this comparison with access to both robotic and linear accelerator radiosurgery techniques as well as research methodology expertise in clinical trials technology assessment, and health services research.

ELIGIBILITY:
Inclusion Criteria:

* 1-3 brain metastases from a confirmed primary extra-cranial site

Exclusion Criteria:

* Any brain metastasis >3cm in maximal diameter
* Easter Cooperative Oncology Group (ECOG) performance status >2
* Prior surgical resection or radiosurgery of a brain metastasis
* Lesion causing significant mass effect (>1cm midline shift)
* Lesion located <5mm from optic chiasm or within the brainstem
* Requires more than one fraction of radiosurgery
* Primary disease histology unknown, lymphoma or germ cell tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Radiosurgery planning and delivery time | 14 days
  Radiosurgery Planning Time: 1) Immobilization Device Fitting 2) CT Simulation and Data Aquisition 3) Treatment Planning 4) Quality Assurance
  Treatment Delivery Time: 1) Patient Setup 2) Target Localization 3) Plan Delivery

SECONDARY OUTCOMES:
Local Control | One Year
  Local Control will be assesed using contrast enhanced MRI at 3,6 and 12 months after radiosurgery
Scattered Radiation Dose | 14 Days
  Thermo-luminescent dosimeters will be placed on the patient during treatment delivery to measure scatter radiation dose
Quality of Life | One Year
  EQ-5D testing will be done prior to radiosurgery and at 4 weeks and at 3,6 and 12 months after radiosurgery
Dosimetry | 7 Days
  Once the plan is approved all dosimetric measures will be recorded.
Acute Toxicity | 3 months
  NCI Common Terminology Criteria for Adverse Events Version 4 will be used to assess acute toxicity up to and including the 3 month post radiosurgery visit
Late Toxicity | One Year
  NCI Common Terminology Criteria for Adverse Events version 4 will be used to assess late toxicity from the 3 month visit to the 12 month visit.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whelan, MD FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Boudreau R, Clark M, Nkansah E. TomoTherapy, GammaKnife and CyberKnife Therapies for Patients with Tumours of the Lung, Central Nervous System, or Intra-abdomen: A Systematic Review of Clinical Effectiveness and Cost Effectiveness. Ottawa: Canadian Agency for Drugs and Technologies in Health; 2009.
- [Background] Gaspar LE, Mehta MP, Patchell RA, Burri SH, Robinson PD, Morris RE, Ammirati M, Andrews DW, Asher AL, Cobbs CS, Kondziolka D, Linskey ME, Loeffler JS, McDermott M, Mikkelsen T, Olson JJ, Paleologos NA, Ryken TC, Kalkanis SN. The role of whole brain radiation therapy in the management of newly diagnosed brain metastases: a systematic review and evidence-based clinical practice guideline. J Neurooncol. 2010 Jan;96(1):17-32. doi: 10.1007/s11060-009-0060-9. Epub 2009 Dec 4. PMID 19960231
- [Result] Regis J, Tamura M, Guillot C, Yomo S, Muraciolle X, Nagaje M, Arka Y, Porcheron D. Radiosurgery with the world's first fully robotized Leksell Gamma Knife PerfeXion in clinical use: a 200-patient prospective, randomized, controlled comparison with the Gamma Knife 4C. Neurosurgery. 2009 Feb;64(2):346-55; discussion 355-6. doi: 10.1227/01.NEU.0000337578.00814.75. PMID 19190462
- [Result] Wowra B, Muacevic A, Tonn JC. Quality of radiosurgery for single brain metastases with respect to treatment technology: a matched-pair analysis. J Neurooncol. 2009 Aug;94(1):69-77. doi: 10.1007/s11060-009-9802-y. Epub 2009 Feb 1. PMID 19184641
- [Result] Blonigen BJ, Steinmetz RD, Levin L, Lamba MA, Warnick RE, Breneman JC. Irradiated volume as a predictor of brain radionecrosis after linear accelerator stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):996-1001. doi: 10.1016/j.ijrobp.2009.06.006. Epub 2009 Sep 23. PMID 19783374
- [Result] Gwak HS, Yoo HJ, Youn SM, Lee DH, Kim MS, Rhee CH. Radiosurgery for recurrent brain metastases after whole-brain radiotherapy : factors affecting radiation-induced neurological dysfunction. J Korean Neurosurg Soc. 2009 May;45(5):275-83. doi: 10.3340/jkns.2009.45.5.275. Epub 2009 May 31. PMID 19516944
- [Result] Chang EL, Hassenbusch SJ 3rd, Shiu AS, Lang FF, Allen PK, Sawaya R, Maor MH. The role of tumor size in the radiosurgical management of patients with ambiguous brain metastases. Neurosurgery. 2003 Aug;53(2):272-80; discussion 280-1. doi: 10.1227/01.neu.0000073546.61154.9a. PMID 12925241
- See also: Robotic Radiosurgery System — http://www.cyberknife.com
- See also: Fixed Gantry Radiosurgery System — http://www.varian.com